CLINICAL TRIAL: NCT01477801
Title: Effects of Cholecalciferol Supplementation in Patients With Chronic Heart Failure and LOw vITamind D Levels. A Phase 2 Randomized Double Blind Study
Brief Title: Effects of Cholecalciferol Supplementation in Patients With Chronic Heart Failure and LOw vITamind D Levels
Acronym: ECSPLOIT -D
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Unita' Sanitaria Locale Di Modena (Other)
Collaborators: Abiogen Pharma (Industry)
Responsible Party: Principal Investigator, TURRINI FABRIZIO, MD, Azienda Unita' Sanitaria Locale Di Modena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCV-MO-11-001; 2011-001726-14 (EudraCT Number)
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Heart Failure; Vitamin D Deficiency
MeSH Terms: conditions — Heart Failure; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHOLECALCIFEROL (Experimental)
  Interventions: Drug: CHOLECALCIFEROL
- PLACEBO (Placebo Comparator)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: CHOLECALCIFEROL — Standard guideline based therapy plus cholecalciferol:
  Loading dose 300.000 U then 50.000 U every month for six months
  Other Names: DIBASE (ABIOGEN PHARMA)
  Arms: CHOLECALCIFEROL
Drug: PLACEBO — Standard guideline based therapy plus placebo
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to determine whether cholecalciferol supplementation in patients with chronic heart failure and low vitamin D levels improves:

1. performance at six minutes walking test
2. echocardiographic parameters
3. neurohormonal imbalance

ELIGIBILITY:
Inclusion Criteria:

* Heart failure diagnosis according to European Society of Cardiology Guideline criteria
* Age > 60 years old
* 25(OH) Vitamin D level < 30 ng/ml
* Clinical and therapeutic stability for one month (NYHA class II or III)

Exclusion Criteria:

* Chronic use of anticonvulsants or barbiturates, steroids, thiazides, aluminium or magnesium, colestipol or cholestyramine
* Glomerular filtration rate lower than 30 ml/min/1.73 m2 according to MDRD equation
* Nephrolitiasis, Sarcoidosis or hypercalcemia
* Recent (three months) acute coronary syndrome or stroke or major vascular surgery
* Reduced life expectancy due to other diseases (active neoplasms, liver cirrhosis...)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
SIX MINUTE WALKING TEST DISTANCE | six months

SECONDARY OUTCOMES:
ECHOCARDIOGRAPHIC PARAMETERS | six months
NEUROHORMONAL CHANGES | six months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Turrini, MD, Principal Investigator — Azienda USL di Modena; Marco Bondi, MD, Study Director — Azienda USL di Modena; Paola Loria, MD, Study Chair — Università di Modena
Locations (1):
- Medicina Cardiovascolare - NOCSAE - Azienda USL, Modena, (mo), Italy